CLINICAL TRIAL: NCT06197178
Title: A Phase 1, Open-Label Study Evaluating the Safety, Tolerability and Efficacy of (LCAR)-G08, a Chimeric Antigen Receptor (CAR)-T Cell Therapy Targeting Guanylyl Cyclase C (GCC) in Subjects With Advanced Gastrointestinal Tumors
Brief Title: A Study of LCAR-G08 in Subjects With Advanced Gastrointestinal Tumors Expressing Guanylyl Cyclase C (GCC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: achieved the proof of concept
Sponsor: Peking University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2301-0001
Record Dates: First submitted 2023-11-20; First posted 2024-01-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2024-12

CONDITIONS: Advanced Gastrointestinal Tumors
Keywords: Advanced Gastrointestinal Tumors

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric Antigen Receptor T cell LCAR-G08 Cells (Experimental): Each subject will receive LCAR-G08 Cells
  Interventions: Biological: LCAR-G08 cells

INTERVENTIONS:
Biological: LCAR-G08 cells — Prior to infusion of the LCAR-G08, subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine.

SUMMARY:
This is a phase 1, single-arm, open-label, dose escalation and expansion study of LCAR-G08 in adult subjects with advanced gastrointestinal tumors expressing guanylyl cyclase C (GCC).

DETAILED DESCRIPTION:
This is a phase 1, single-arm, open-label, dose escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy profiles of the cell-based LCAR- G08 in subjects with guanylyl cyclase C (GCC)-positive advanced gastrointestinal tumors. Subjects who meet the eligibility criteria will receive LCAR-G08 infusion. The study will include the following sequential phases: screening, pre-treatment (cell product preparation; lymphodepleting chemotherapy), treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Histologically confirmed metastatic colorectal cancers and other advanced gastrointestinal cancers (esophageal cancer, gastric cancer, pancreatic cancer, and small bowel cancer).
* Aged 18 to 70 years, either sex.
* GCC immunohistochemistry (IHC) staining is positive.
* At least one measurable tumor lesion according to RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Expected survival ≥ 3 months.
* Clinical laboratory values meet screening visit criteria.

Exclusion Criteria:

* Previous CAR-T cell, T cell receptor-engineered (TCR) T cell, or therapeutic tumor vaccination treatment within the past 6 months; and the corresponding CAR-T, TCR-T cells can still be detected.
* Ever received any treatment targeting GCC.
* Prior antitumor therapy with insufficient washout period.
* Brain metastases.
* Pregnant or lactating women.
* Hepatitis C virus (HCV) antibody-positive or human immunodeficiency virus (HIV) antibody-positive, active syphilis, Epstein-Barr virus (EBV) infected.
* Severe underlying disease.
* Presence of other serious pre-existing medical conditions that may limit patient participation in the study.Any condition that, in the investigator's judgment, will make the subject unsuitable for participation in this study.

Any condition that, in the investigator's judgment, will make the subject unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate | Minimum 2 years after LCAR-G08 infusion (Day 1)
  Dose-limiting toxicity (DLT) refers to a drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose.
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Minimum 2 years after LCAR-G08 infusion (Day 1)
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment.
Recommended Phase 2 Dose (RP2D) regimen finding | Minimum 2 years after LCAR-G08 infusion (Day 1)
  RP2D established through accelerated titration design (ATD) and Bayesian Optimal Interval (BOIN) design.
Maximum concentration (Cmax) | Minimum 2 years after LCAR-G08 infusion (Day 1)
  The maximum observed concentration of CAR positive T cells or transgene CAR copy number after LCAR-G08 infusion.
Time to Cmax (Tmax) | Minimum 2 years after LCAR-G08 infusion (Day 1)
  The time it takes to reach the maximum concentration or time to Cmax after LCAR-G08 infusion.
Time to the last observed concentration | Minimum 2 years after LCAR-G08 infusion (Day 1)
  The time it takes to reach the last observed concentration after LCAR-G08 infusion.
Area Under the Curve (AUC) last | Minimum 2 years after LCAR-G08 infusion (Day 1)
  The total exposure of the drug experienced by the subject in a clinical study from LCAR-G08 infusion to time to the last observed concentration.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) after administration | Minimum 2 years after LCAR-G08 infusion (Day 1)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve complete response (CR) or partial response (PR) after treatment via LCAR-G08 cell infusion, and the objective tumor response rate will be calculated for patients with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 only.
Disease Control Rate (DCR) after administration | Minimum 2 years after LCAR-G08 infusion (Day 1)
  Disease Control Rate (DCR) is defined as the proportion of patients with complete response, partial response and stable disease.
Duration of Remission (DoR) after administration | Minimum 2 years after LCAR-G08 infusion (Day 1)
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (PR or better) to the first documented disease progression evidence (according to RECIST 1.1) of the responders (who achieve PR or better response).se).
Time to Response (TTR) after administration | Minimum 2 years after LCAR-G08 infusion (Day 1)
  Time to Response (TTR) is defined as the time from the date of first infusion of LCAR-G08 to the date of the first response evaluation of the subject who has met all criteria for PR or better.
Progression-free Survival (PFS) after administration | Minimum 2 years after LCAR-G08 infusion (Day 1)
  Progression-free Survival (PFS) is defined as the time from the date of first infusion of the LCAR-G08 to the first documented disease progression (according to RECIST 1.1) or death (due to any cause), whichever occurs first.
Overall Survival (OS) after administration | Minimum 2 years after LCAR-G08 infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LCAR-G08 to death of the subject.
Incidence of anti-LCAR-G08 antibody and positive sample titer | Minimum 2 years after LCAR-G08 infusion (Day 1)
  Venous blood samples will be collected to measure LCAR-G08 positive cell concentrations and the transgenic level of LCAR-G08, at the time points when anti-LCAR-G08 antibody serum samples are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital & Institute, Beijing, Beijing Municipality
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No